CLINICAL TRIAL: NCT06958510
Title: Modified Anatomical Mesh In The Management Of Orbito-Zygomatico-Maxillary Complex Fractures. A Randomized Clinical Trial
Brief Title: Modified Anatomical Mesh In The Management Of Orbito-Zygomatico-Maxillary Complex Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3D-MAM
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-04

CONDITIONS: Orbital Fractures; Zygomatic Fractures
Keywords: anatomical mesh; 3D-mesh; orbital mesh; orbital fracture; zygomatic fracture; reconstruction
MeSH Terms: conditions — Orbital Fractures; Zygomatic Fractures

STUDY DESIGN:
Intervention Model Description: Patients with Orbito-Zygomaticomaxillary complex fractures with orbital floor defect managed with 3D-Modified Anatomic Mesh
Who Masked: Participant
Masking Description: Sequentially numbered, opaque, sealed envelopes (SNOSE) allocation concealment method will be utilized. Each participant included in the study will be given a serial number that will be used in the allocation. These numbers will be written in identical sheets of paper with the group to which each participant is allocated and placed inside opaque envelopes carrying the respective names of participants. A trial independent personnel will be assigned the role of keeping the envelopes and unfolding them only at the time of the operation, so that the participant is allocated to a group which is concealed from the operator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Orbito-Zygomaticomaxillary Complex fracture managed with 3D-Modified Anatomical-Mesh (Active Comparator): Patients with Orbito-Zygomaticomaxillary Complex fracture managed with 3D-Modified Anatomical-Mesh
  Interventions: Device: 3D-Modified Anatomical-Mesh.
- Patients with Orbito-Zygomaticomaxillary Complex fracture managed with conventional orbital rim mini (Experimental): Patients with Orbito-Zygomaticomaxillary Complex fracture managed with conventional orbital rim mini
  Interventions: Device: conventional orbital rim miniplates and orbital mesh configuration

INTERVENTIONS:
Device: 3D-Modified Anatomical-Mesh. — 3D-Modified Anatomical-Mesh.
  Arms: Patients with Orbito-Zygomaticomaxillary Complex fracture managed with 3D-Modified Anatomical-Mesh
Device: conventional orbital rim miniplates and orbital mesh configuration — conventional orbital rim miniplates and orbital mesh configuration
  Arms: Patients with Orbito-Zygomaticomaxillary Complex fracture managed with conventional orbital rim mini

SUMMARY:
Orbito-Zygomaticomaxillary-complex fractures is a form of a complex orbital floor fracture, with affection of the inferior orbital rim and the orbital walls. According to published research, between 67 - 84 % of periorbital bone fractures are orbital floor fractures.

Evaluation of 3D-Modified Anatomic Mesh in the management of OZM- complex fractures with orbital floor defect, and compare it with the conventional fixation configuration.

DETAILED DESCRIPTION:
Patients suffering from OZM- complex fractures was treated using 3D-Modified Anatomical Mesh for orbital floor reconstruction and orbital rim fixation. Patients was randomly allocated into study and control groups, where it is managed with the conventional 2.0-miniplate and stock mesh. A standardized surgical protocol was followed in both groups. Patients was clinically evaluated for pain, wound healing, nerve sensation, ocular motility and diplopia, and tarsal plate morphology. Moreover, radiographic survey was performed post operatively to assess the proper positioning of the implant, to confirm proper fracture reduction, and radiographic enophthalmos analysis

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from Orbito-Zygomaticomaxillary complex fractures with fracture in the orbital floor and orbital floor defect(16).
2. Fractures that are indicated for open reduction and internal fixation.
3. Patients suffering from ocular complications:

   1. Monocular diplopia.
   2. Enophthalmos above 2 mm.
   3. Restricted ocular motility.
4. Patients with orbital wall defects with orbital soft tissue herniation into the maxillary sinus.
5. Adult patient either male or female that agrees to present for follow-up visits for an adequate postoperative period.

Exclusion Criteria:

1. Patients with isolated orbital floor defects and blowout fractures.
2. Patients with isolated zygomatico-maxillary complex fracture with no orbital floor/ walls defects.
3. Patients with bilateral orbital defects.
4. Patients with Infected wounds in periorbital region.
5. Medically compromised patients rendering them inoperable.
6. Patients with ruptured globe or blindness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Radiographic assessment of the management of the Orbito-Zygomaticomaxillary Complex fracture | 1 week
  Radiographic assessment of the management of the Orbito-Zygomaticomaxillary Complex fracture

SECONDARY OUTCOMES:
Periorbital ecchymosis | 6 weeks
  Postoperative periorbital ecchymosis will be evaluated on a 3-points scale (0-3). The scoring system divides ecchymosis into upper and lower eyelids, and furthermore into thirds for each eyelid.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP
Access Criteria: to any one who required them after deidentification